CLINICAL TRIAL: NCT03876730
Title: Assessment of the Use of Lower Extremity Orthosis in Children With Cerebral Palsy Within The Scope of International Classification of Functioning, Disability and Health
Brief Title: International Classification of Functioning, Disability and Health and Lower Extremity Orthoses in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sefa Üneş, Priciple Investigator, Hacettepe University
Other Study IDs: Sefaunes
Record Dates: First submitted 2019-02-08; First posted 2019-03-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Lower Extremity Orthosis; ICF Core Set
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 3-18 aged children with cerebral palsy
  Interventions: Other: ICF CP Core Set

INTERVENTIONS:
Other: ICF CP Core Set — Core set

SUMMARY:
International Classification of Functioning, Disability and Health (ICF) is a coding system developed to describe the health status of individuals in a universal way. The increasingly common core sets are short forms of ICF categories that are specifically selected for diseases. The aim of this study is to investigate the relationship among the lower extremity orthoses commonly used in children with cerebral palsy (CP), body structure and functions, activity and participation level, and is to determine the relationship between clinical tests and ICF CP core set. For this purpose, a total of 75 children with ages between 3 and 18 will be divided into 3 groups, including using a walking orthosis, using a resting orthosis, and using both walking and resting orthoses. Children's muscle tone, joint limitation, gross motor functions, balance skills, activity and participation levels and quality of life will be assessed with the tests frequently used in the clinic separately and with the core set in a holistic framework.

ELIGIBILITY:
Inclusion Criteria:

* Being 3-18 age years old
* Having the diagnosis with cerebral palsy
* Being no Botulinum Toxin Application or no surgery for the last 6 months

Exclusion Criteria:

* If there is any other neurological or orthopedic problem other than cerebral palsy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The children who will come to the investigator's unit, Cerebral Palsy and Pediatric Rehabilitation
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale (PBS) | 3 minutes
  PBS is a 14-item scale that assesses children's balance. Each item is scored between 0 and 4 points. As a result, the total score is given, while the low score refers to the poor balance and the high score refers to the good balance.
Gross Motor Function Measurement (GMFM)-88 | 5 minutes
  Children's motor ability will be assessed to investigate the correlations between the motor functions and orthosis used by child. The GMFM-88 consists of 88 items examining children's gross motor movements. Each item is scored between 0 and 3 points. The higher the child gets, the more successful the child is in gross motor functions.
Measurements of range of motions | 5 minutes
  Goniometer will be used to determine the range of motions. So, the investigators will be able to investigate the correlations between orthotic and joints
Modified Ashworth Scale (MAS) | 5 minutes
  MAS will be used to determine the muscle tone. MAS is a scale that shows muscle hypertone between 0 and 5. 5 means that the joint is rigid due to the increase in excess tonus while 0 means no increase in tonus.
Pediatric Quality of Life (PedsQL) | 5 minutes
  PedsQL is a quality-of-life questionnaire which evaluates the situations encountered in daily life of children with CP such as dressing, self-care, school activities, speech and eating. Special PedsQL will be used in 4 different age groups, including 3-4 age specific, 5-7 age specific, 8-12 age specific and 13-18 age specific. The number of items in each age group is different, but the result of PedsQL is expressed in%, not total points. A higher score refers to a more independent child.
Pediatric Functional Independence Measurement (WeeFIM) | 5 minutes
  WeeFIM is an 18-item scale that measures children's activity and participation. It consists of 18 items including self-care, sphincter control, locomotion, memory, etc. Each item is scored between 0 and 7. A higher score refers to a more independent child.

SECONDARY OUTCOMES:
ICF CP Core Set | 10 minutes
  CP Core set consists of totally 25 items about body functions, body structure, activity, participation and environmental factors. Each item is scored within 0 to 4 points. 0 indicates that there are no problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No